CLINICAL TRIAL: NCT06124482
Title: Performance and Safety Evaluation of the FHK®-CK Knee Prosthesis Indicated for the Treatment of Primary and Secondary First Line Gonarthrosis and Revision Arthroplasty - 2 Years Follow-up - A Pilot Study
Brief Title: Performance and Safety Evaluation of the FHK®-CK Knee Prosthesis
Acronym: FHK-CK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FH ORTHO (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-01
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Complex primary Total Knee Arthroplasty; Revision Total Knee Arthroplasty; Functional performance; Safety evaluation
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Two target populations will be included in this clinical investigation :
  * 60 patients requiring primary Total Knee Arthroplasty
  * 32 patients requiring revision Knee Arthroplasty.
  In this clinical investigation, it was not possible to realize a double-blinding for practical reasons. Nevertheless, a collection of the primary outcome (score KSS) will be realized blindly to the surgeon in charge of the patient by an intervener not involved in the medical care of the patient, who did not participate in the intervention and did not collect the preoperative KSS score.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Knee replacement (Experimental): Implantation of FHK-CK prosthesis either for a complex primary arthroplasty or for revision intend
  Interventions: Device: Total Knee arthroplasty

INTERVENTIONS:
Device: Total Knee arthroplasty — The FHK-CK prosthesis (non CE-Marked, class III) is to be implanted with the use of FHK-CK instruments. The surgery has to be performed in accordance with the practice/guidelines, FHK-CK Instruction For Use (IFU) and surgical techniques documents.

SUMMARY:
The life expectancy worldwide is increasing and leading to an increase of knee arthroplasty. Also, as millions of people around the world are currently living with a Total Knee Arthroplasty (TKA), the need for revision surgery represents a large public health burden. In this context, FH ORTHO company develops FHK®-CK (prosthesis + ancillary equipment) which is a knee prosthesis for complex first intention and revision knee arthroplasty. This new medical device complements the FHK® standard first-line range (CE marked).

The FHK®-CK ancillary equipment were designed by expert knee surgeons and is simple, reliable and reproducible. It allows for maximum versatility while remaining compact.

By completing the FHK® range of first intention prostheses, the FHK®-CK allows the surgeon to be on the same level as the competitors by having a first intention and semi-constrained prosthesis. This prosthetic arsenal allows the surgeon to opt for the best solution for his patient so that he can regain mobility and a satisfactory quality of life. Also, in case of failure of the FHK® first-line prosthesis, it will provide the surgeon and the patient with a simple alternative to prosthesis replacement. As it has been developed in line with the first intention, inter-compatibility between the two systems is possible, which simplifies the surgical procedure and reduces the risks for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring knee arthroplasty for primary or secondary gonarthrosis:

  * For primary intention arthroplasty: Patient with either
  * major axial deviation,
  * major peripheral failure or
  * bone defect;

    * For prosthesis revision surgery: Patient who have had a failed 1st implantation, with or without bone defects.
* Patient able to understand and answer the questionnaires provided by the protocol;
* Subject affiliated to a health insurance system or is a beneficiary;
* Signed informed consent form (ICF) for participation to the research.

Exclusion Criteria:

* Patient with an ongoing acute infection, outside knee to be operated;
* Patient with a mental or neuromuscular disorder that would create an unacceptable risk of prosthetic instability, prosthetic fixation failure or post-operative complications;
* Patient with a known allergy to any of the components of the FHK®-CK implants (Nickel, Cobalt, Chromium);
* Patient with a dependency (drug, alcohol,…) that could affect his/ her ability to comply with the protocol, at the investigator's discretion;
* Patient requiring knee reconstruction;
* Patient with any medically significant findings or significant history that may impact the safety, interpretation of results, and/ or participation of the subject in the clinical trial, as determined by the investigator;
* Patient with an existing knee or hip prosthesis (outside knee to be operated) that may impact the evaluation of the FHK®-CK prosthesis;
* Patient concurrently participating in another clinical trial or who has recently participated in another clinical trial for which the exclusion period has not been completed.
* Vulnerable subjects :

  * Pregnant, parturient, or breastfeeding women,
  * Subject deprived of liberty, hospitalized without consent or admitted to a health or social establishment for purposes other than that of research,
  * Minor,
  * Adult under protective supervision (tutorship, curatorship),
  * Subject not able to understand the subject information leaflet (e.g. for linguistic or psychiatric reasons) and/or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Functional performance | Baseline (preoperatively), at 6 weeks, 6 months, 12 months and 24 months after surgery.
  Evolution of the functional performance of FHK®-CK prosthesis using the KSS scoring system, which is composed of 2 sections : Knee score (KSKS) and function score (KSFS). Each section is scored on a scale of 0 to 100 ; the higher the score, the better the overall functionality of the knee. The functional performance of the FHK®-CK prosthesis will be demonstrated at 2 years if an improvement of the KSKS and KSFS scores at least equal to the Minimal Clinically Important Difference (MCID) values is observed.

SECONDARY OUTCOMES:
Adverse and serious adverse events evaluation | Through study completion, an average of 2 years
  Occurrence of adverse and serious adverse events, including complication
Revision rate evaluation | At 6 weeks, 6 months, 12 months and 24 months after surgery.
  Revision rate
Evaluation of patient's tolerance of the FHK-CK prosthesis | At 6 weeks, 6 months, 12 months and 24 months after surgery.
  Tolerance assessed by the surgeon with a 4-Likert scale (very bad - bad - good - very good)
Device deficiencies evaluation | Through study completion, an average of 2 years
  Number of device deficiencies and description of deficiencies.
Quality of life assessment | Baseline (preoperatively), at 6 months, 12 months and 24 months after surgery.
  Self assessement of quality of life using the medical outcome study Short Form (SF-12) scale (General Quality of life score) from 0 "worst quality of life" to 100 "best quality of life".
Quality of life assessment | Baseline (preoperatively), at 6 months, 12 months and 24 months after surgery.
  Self assessement of quality of life using the Oxford Knee score (OKS), especially developed for knee surgery. The OKS is derived from 12 questions assessed on a Likert scale with values from 0 to 4; a summative score is then calculated where 48 is the best possible score (least symptomatic) and 0 is the worst possible score (most symptomatic)
Patient's satisfaction about FHK®-CK prosthesis | At 6 months, 12 months and 24 months after surgery
  Satisfaction assessed by the patient with a 4-Likert scale ((very bad - bad - good - very good)
Surgeon's satisfaction about FHK®-CK equipment | During surgery
  Satisfaction assessed by the surgeon for each surgery performed with FHK®-CK with a specific questionnaire developed including 9 questions with either a lickert scale or a yes/no response.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Privé La Châtaigneraie, Beaumont
  - CHRU de la Cavale Blanche, Brest
  - Hôpital Beaujon AP-HP, Clichy
  - Hôpital Raymond Poincaré AP-HP, Garches
  - CH d'Haguenau, Haguenau
  - Centre Hospitalier Régional Universitaire de Nancy, Nancy
  - Groupe Hospitalier Pitié Salpêtrière AP-HP, Paris